CLINICAL TRIAL: NCT01464528
Title: Use Of Hyaluronic Acid Gel To Prevent Intrauterine Adhesions In Hysteroscopic Surgery
Brief Title: Safety Study of Use of Hyaluronic Acid Gel To Prevent Intrauterine Adhesions In Hysteroscopic Surgery
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HYALOBARRIER- HMO-CTIL
Record Dates: First submitted 2011-08-15; First posted 2011-11-03 (Estimated); Last update posted 2011-11-03 (Estimated); Status verified 2011-07

CONDITIONS: Tissue Adhesions
Keywords: hysteroscopy; postoperative complications; adhesions; hyaluronic gel; prevention
MeSH Terms: conditions — Tissue Adhesions; Postoperative Complications | interventions — Hyaluronic Acid; Ethanol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Hyaluronan (Active Comparator): Use of hyaluronic acid gel
  Interventions: Drug: Hyaluronan
- control (No Intervention)

INTERVENTIONS:
Drug: Hyaluronan — single use of 10 mL of the hyalobarrier gel intrauterine immediately following hysteroscopic surgery
  Other Names: hyaluronic acid, alcohol and carboxil
  Arms: Hyaluronan

SUMMARY:
Operations in the uterus are currently possible using a hysteroscope. One serious though rare complication of such procedures is the development of intra-uterine adhesions. There currently are no methods to prevent this. The aim of this study is to evaluate the safety of using hyaluronic gel after hysteroscopic surgery.

DETAILED DESCRIPTION:
Operations in the uterus are currently possible using a hysteroscopic approach. Intrauterine procedures include; polypectomy, myomectomy, removal of lost IUD,removal of a septum and more. One serious though rare complication of operative hysteroscopy is the development of intra-uterine adhesions. Such adhesions, also known as asherman's syndrome, can cause serious consequences such as infertility and miscarriage. The hypothesis is that the removal of the endometrium and the exposure of ra uterine wall to each other can cause attachment and adhesions. the treatment is to mechanically break the adhesion. recurrence is however common. There currently are no methods to prevent adhesions following curettage or hysteroscopy. The aim of this study is to evaluate the safety of using hyaluronic gel after hysteroscopic surgery. At a later research, the efficacy of barrier gel will be measures.

ELIGIBILITY:
Inclusion Criteria:

* age 18 year old and over
* need of hysteroscopic surgery

Exclusion Criteria:

* preoperative fever or infection
* malignancy
* previous PID
* contraindications for anesthesia
* pregnancy
* under 18 year old
* not able to read and/or understand informed consent
* taking any medicine other than oral contraceptives

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2011-11; Primary Completion 2012-03 (Estimated); Study Completion 2012-05 (Estimated)

PRIMARY OUTCOMES:
Patient satisfaction following gel application | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Ariel Revel, MD, Principal Investigator — Hadassah